CLINICAL TRIAL: NCT02990923
Title: The Effect of High-Flow Needleless Valve and DualCap Disinfection Devices on Incidence of Catheter-related Bloodstream Infection in Hemodialysis Patients: a Single Center Randomized Controlled Trial
Brief Title: High-Flow Needleless Valve and DualCap Disinfection Devices Associate With Catheter-related Bloodstream Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Rong Xu, vice professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PekingHDNC
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Catheter-related Bloodstream Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): In this group, patients will use traditional standard hemodialysis connector and receive typical disinfection management
- Only High-Flow Valve (Experimental): In this group, patients will use High-Flow Needleless Valve instead of traditional standard hemodialysia connector, but still receiving typical disinfection management
  Interventions: Device: High-Flow Needleless Valve
- Both Divices (Experimental): In this group, patients will receive both High-Flow Needleless Valve and DualCap Disinfection Devices in hemodialysis
  Interventions: Device: High-Flow Needleless Valve; Device: DualCap Disinfection Devices

INTERVENTIONS:
Device: High-Flow Needleless Valve
  Arms: Both Divices; Only High-Flow Valve
Device: DualCap Disinfection Devices
  Arms: Both Divices

SUMMARY:
The purpose of this study is to investigate whether the usage of High-Flow Needleless Valve and DualCap Disinfection Devices would reduce the incidence of catheter-related bloodstream infection in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Implanted non-tunneled cuff catheter for any reason and going on blood purified therapy in our centre
* Have signed information consent form

Exclusion Criteria:

* Have got bacteremia before catheter implantation
* Catheter changing in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Catheter-related bloodstream infection | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Number of participants with catheter withdraw for any reason | through study completion, an average of 1 year
Number of participants with catheter dysfunction | through study completion, an average of 1 year